CLINICAL TRIAL: NCT01787461
Title: Randomized, Double-blind, Placebo Controlled Trial Assessing The Effects Of An Oral Dietary Supplement Containing Marine And Plant Extracts On Overall Facial Skin Appearance Among Healthy Adult Women With Photo-aged Skin
Brief Title: A Study to Assess the Effects of an Oral Dietary Supplement on Overall Facial Appearance Among Healthy Adult Women With Existing Skin Damage From Sun Exposure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B5271003
Record Dates: First submitted 2012-12-05; First posted 2013-02-08 (Estimated); Results first posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Photodamaged Skin
Keywords: Trial assessing effects of an oral dietary supplement on overall facial appearance among healthy women with photodamaged skin.
MeSH Terms: interventions — Imedeen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imedeen (Experimental): Imedeen is the study product
  Interventions: Dietary Supplement: Imedeen
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Imedeen — Two tablets per day for 6 months
  Other Names: Imedeen Time Perfection
  Arms: Imedeen
Dietary Supplement: Placebo — Two tablets per day for 6 months
  Arms: Placebo

SUMMARY:
The study hypothesis is that Imedeen will show effects on skin health, when compared to placebo over a 6 month intervention period with respect to changes in skin appearance, skin density, moisture, and in fine lines and wrinkles.

ELIGIBILITY:
Inclusion Criteria:

In general good health and have no contraindications to the study product; Have Fitzpatrick Skin Type I-IV as determined by a trained evaluator. Have Glogau Classification of Photoaging of II or III as determined by the investigator.

Exclusion Criteria:

Use of any dietary supplement, over-the-counter or prescription product with the indication of improving the appearance or condition of the skin within one month of baseline.

History of or current disease or condition of the skin that the investigator deems inappropriate for participation (eg, atopic skin, facial scars, psoriasis, eczema, other scaly inflammatory diseases).

Subjects who have had a facial cosmetic procedures (eg, fillers, toxins, facial peel) or invasive surgical procedures (eg, laser treatment or face lift) or other facial treatments by a physician or skin care professional within the last 6 to 9 months from baseline (pending procedure type) or plan to have a treatment during the study.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - TKL Research, Inc., Fair Lawn, New Jersey
  - The Education & Research Foundation, Inc., Lynchburg, Virginia
  - McDaniel Institute of Anti-Aging Research, Virginia Beach, Virginia

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5271003&StudyName=A%20study%20to%20assess%20the%20effects%20of%20an%20oral%20dietary%20supplement%20on%20overall%20facial%20appearance%20among%20healthy%20adult%20women%20with%20existing%20ski

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Two Placebo tablets matched to Imedeen, orally daily for 24 weeks.
- Imedeen: Imedeen (two tablets) containing marine complex at 210 (milligrams) mg, vitamin C at 48 mg, zinc at 3.6 g and tomato fruit and grape extract blend at 56 mg, orally daily for 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Imedeen
Started | 96 | 98
Completed | 82 | 89
Not Completed | 14 | 9
Not completed — Adverse Event | 4 | 3
Not completed — Lost to Follow-up | 3 | 2
Not completed — No longer met eligibility criteria | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least one dose of the study treatments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Imedeen | Total
Number analyzed (Participants) | 95 | 98 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (7.38) | 52.7 (6.58) | 52.6 (6.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 98 | 193
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Investigator Global Assessment (IGA) of Participant's Overall Facial Appearance at Week 24
Description: IGA of overall facial appearance was measured using a numerical severity rating scale of 0 to 9 using 1/2 points, where 0 to less than or equal to (<=) 3 signifies Mild; greater than (>) 3 to <=6 signifies Moderate and >6 to <=9 signifies Severe.
Time Frame: Baseline, Week 24
Population: Modified intent-to-treat (m-ITT) population included all randomized participants who had at least 1 pre-dose and post-dose assessment value. Here "n" signifies those participants who were evaluable for this measure at specified time- points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
units on scale
  Baseline (n=93,97) | 6.04 (1.45) | 5.81 (1.30)
  Change at Week 24 (n=92,95) | 0.6 (1.28) | 0.7 (1.23)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Change at Week 24: Analysis was performed using an analysis of variance (ANOVA) model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.358, ANOVA; Least Squares (LS) Mean Difference = 0.14, 95% CI 2-sided [-0.16 to 0.44]

2. Secondary Outcome: Photographic Assessment Compared to Baseline of the Participants Overall Facial Appearance by Independent Panel Review Committee (IPRC) at Week 24
Description: IPRC assessment was performed in accordance with the Canfield procedures and rated the improvement relative to Baseline. The investigators used an improvement scale that ranged from -3 to 3 (where -3 = Definite worsening, -2 = Moderate worsening, -1 = Slight worsening, 0 = No change, 1 = Slight improvement, 2 = Moderate improvement, 3 = Definite improvement).
Time Frame: Week 24
Population: m-ITT population included all randomized participants who had at least 1 pre-dose and post-dose assessment value. Here "N" (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 94
units on scale | -0.2 (0.86) | -0.1 (0.82)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Analysis was performed using Cochran-Mantel-Haenszel (CMH) test with modified ridit scores, controlling for Glogau classification of photoaging and site; Test type: Superiority or Other; p = 0.568, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.037, 95% CI 2-sided [-0.19 to 0.27]

3. Secondary Outcome: Change From Baseline in Investigator Global Assessment (IGA) of Participant's Overall Facial Appearance at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: m-ITT population included all randomized participants who had at least 1 pre-dose and post-dose assessment value. Here "n" signifies those participants who were evaluable for this measure at specified time- points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
units on scale
  Baseline (n=93,97) | 6.04 (1.45) | 5.81 (1.30)
  Change at Week 12 (n=92,95) | 0.4 (1.14) | 0.4 (1.07)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Change at Week 12: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.797, ANOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.25 to 0.33]

4. Secondary Outcome: Change From Baseline in Investigator Assessment of Face at Weeks 12 and 24
Description: Investigator performed the assessment of face (Fine lines/wrinkles (L/W) of the periocular area (A), Fine lines/wrinkles of the perioral area, dark circles (dc) or "bags" under the eye, mottled hyperpigmentation (MH), sallowness/yellowing, roughness/texture) using a numerical severity rating scale of 0 to 9, where 0 to less than or equal to (<=) 3 signifies Mild; greater than (>) 3 to <=6 signifies Moderate and >6 to <=9 signifies Severe.
Time Frame: Baseline, Week 12, 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
units on scale
  Baseline: Fine L/W Periocular A (n=93,97) | 5.95 (1.50) | 5.79 (1.44)
  Baseline: Fine L/W Perioral A (n= 93,97) | 4.89 (1.78) | 4.69 (1.65)
  Baseline: Under eye dc or bags(n= 93,97) | 5.68 (1.55) | 5.34 (1.44)
  Baseline: MH (n=93,97) | 4.95 (1.71) | 5.06 (1.51)
  Baseline: Sallowness/yellowing (n=93,97) | 3.41 (1.42) | 3.51 (1.33)
  Baseline: Roughness/texture (n=93,97) | 3.10 (1.66) | 2.77 (1.50)
  Change at Week 12: Fine L/W Periocular A(n= 92,95) | 0.5 (1.04) | 0.5 (1.09)
  Change at Week 12: Fine L/W Perioral A(n= 92,95) | 0.4 (1.01) | 0.4 (1.07)
  Change at Week 12: Under eye dc or bags (n= 92,95) | 0.5 (1.28) | 0.3 (1.38)
  Change at Week 12: MH (n= 92,95) | 0.3 (1.38) | 0.3 (1.42)
  Change at Week 12: Sallowness/yellowing (n= 92,95) | 0.4 (1.46) | 0.4 (1.45)
  Change at Week 12: Roughness/texture (n= 92,95) | 0.4 (1.63) | 0.2 (1.45)
  Change at Week 24: Fine L/W Periocular A(n= 92,95) | 0.7 (1.31) | 0.8 (1.26)
  Change at Week 24: Fine L/W Perioral A(n= 92,95) | 0.4 (1.14) | 0.5 (1.09)
  Change at Week 24: Under eye dc or bags (n= 92,95) | 0.7 (1.66) | 0.6 (1.37)
  Change at Week 24: MH (n= 92,95) | 0.7 (1.32) | 0.7 (1.36)
  Change at Week 24: Sallowness/yellowing (n= 92,95) | 1.0 (1.43) | 1.0 (1.45)
  Change at Week 24: Roughness/texture (n= 92,95) | 0.8 (1.65) | 0.5 (1.63)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Change at Week 12, Fine lines/wrinkles (Periocular area): Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.965, ANOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.29 to 0.30]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; Change at Week 12, Fine lines/wrinkles (Perioral area): Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.674, ANOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.20 to 0.30]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; Change at Week 12, Under eye dark circles or bags: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.916, ANOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.35 to 0.32]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; Change at Week 12, Mottled hyperpigmentation: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.915, ANOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.39 to 0.35]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; Change at Week 12, Sallowness/yellowing: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.672, ANOVA; LS Mean Difference = -0.07, 95% CI 2-sided [-0.40 to 0.26]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; Change at Week 12, Roughness/texture: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.655, ANOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.27 to 0.43]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; Change at Week 24, Fine lines/wrinkles(Periocular area): Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.561, ANOVA; LS Mean Difference = 0.10, 95% CI 2-sided [-0.23 to 0.43]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; Change at Week 24, Fine lines/wrinkles(Perioral area): Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.356, ANOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.14 to 0.40]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; Change at Week 24, Under eye dark circles or bags: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.669, ANOVA; LS Mean Difference = 0.08, 95% CI 2-sided [-0.28 to 0.43]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; Change at Week 24, Mottled hyperpigmentation: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.954, ANOVA; LS Mean Difference = 0.01, 95% CI 2-sided [-0.32 to 0.34]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; Change at Week 24, Sallowness/yellowing: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.684, ANOVA; LS Mean Difference = -0.06, 95% CI 2-sided [-0.34 to 0.22]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; Change at Week 24, Roughness/texture: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.886, ANOVA; LS Mean Difference = -0.02, 95% CI 2-sided [-0.35 to 0.30]

5. Secondary Outcome: Change From Baseline in Investigator Assessment of Decolletage and Back of Hands at Weeks 12 and 24
Description: Investigator performed the assessment of decolletage and back of hands (crepyness, mottled hyperpigmentation [MH]) using a numerical severity rating scale of 0 to 9 using 1/2 points, where 0 to less than or equal to (<=) 3 signifies Mild; greater than (>) 3 to <=6 signifies Moderate and >6 to <=9 signifies Severe.
Time Frame: Baseline, Week 12, 24
Population: Modified intent-to-treat (m-ITT) population included all randomized participants who had at least 1 pre-dose and post-dose assessment value. Here "n" signifies those participants who were evaluable for this measure at specified time -points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
units on scale
  Baseline: Decolletage-Crepyness (n=93,97) | 4.65 (1.77) | 4.56 (1.60)
  Baseline: Decolletage-MH (n=93,97) | 5.09 (1.80) | 5.08 (1.65)
  Baseline: Back of Hands-Crepyness (n=93,97) | 5.37 (1.43) | 5.19 (1.42)
  Baseline: Back of Hands-MH (n=93,97) | 3.96 (1.53) | 3.92 (1.69)
  Change at Week 12: Decolletage-Crepyness (n=92,95) | 0.2 (1.23) | 0.2 (1.49)
  Change at Week 12: Decolletage-MH (n=92,95) | 0.4 (1.36) | 0.5 (1.20)
  Change at Week 12:Back of Hands-Crepyness(n=92,95) | 0.6 (1.39) | 0.5 (1.48)
  Change at Week 12: Back of Hands-MH (n=92,95) | -0.2 (1.09) | 0.3 (1.08)
  Change at Week 24: Decolletage-Crepyness (n=92,95) | 0.7 (1.56) | 0.7 (1.36)
  Change at Week 24: Decolletage-MH (n=92,95) | 0.6 (1.43) | 0.6 (1.14)
  Change at Week 24:Back of Hands-Crepyness(n=92,95) | 0.7 (1.39) | 0.7 (1.45)
  Change at Week 24: Back of Hands-MH (n=92,95) | 0.1 (1.20) | 0.4 (1.22)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Change at Week 12, Decolletage-Crepyness: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.901, ANOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-0.33 to 0.37]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; Change at Week 12, Decolletage-Mottled Hyperpigmentation: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.399, ANOVA; LS Mean Difference = 0.14, 95% CI 2-sided [-0.19 to 0.47]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; Change at Week 12, Back of Hands-Crepyness: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.875, ANOVA; LS Mean Difference = -0.03, 95% CI 2-sided [-0.38 to 0.32]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; Change at Week 12, Back of Hands-Mottled Hyperpigmentation: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.005, ANOVA; LS Mean Difference = 0.43, 95% CI 2-sided [0.13 to 0.73]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; Change at Week 24, Decolletage-Crepyness: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.876, ANOVA; LS Mean Difference = 0.03, 95% CI 2-sided [-0.33 to 0.38]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; Change at Week 24, Decolletage-Mottled Hyperpigmentation: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.789, ANOVA; LS Mean Difference = 0.05, 95% CI 2-sided [-0.29 to 0.38]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; Change at Week 24, Back of Hands- Crepyness: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.901, ANOVA; LS Mean Difference = 0.04, 95% CI 2-sided [-0.31 to 0.38]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; Change at Week 24, Back of Hands - Mottled Hyperpigmentation: Analysis was performed using an ANOVA model with treatment, Glogau cassification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.027, ANOVA; LS Mean Difference = 0.38, 95% CI 2-sided [0.04 to 0.72]

6. Secondary Outcome: Participants Improvement Assessment of Face at Week 12 and 24
Description: Participants performed the assessment of face (overall facial (OA) appearance, fine lines and wrinkles (L/W) present in the eye area, upper lip, or cheek areas, under eye dark circles (dc) or bags, discoloration [uneven, patchy, blotchy areas of light and dark, age spots, liver spots], complexion/glow [bright radiant appearance] and smoothness) at Baseline using a 10-point numerical scale, and at Week 12, 24 using a 7-point improvement scale. At Baseline, participants rated the facial parameters using a 10-point scale ranging from 1 (Not noticeable) to 10 (Very noticeable). At Week 12 and 24, assessment was performed relative to Baseline using an improvement scale that ranged from -3 to 3 (where -3 = Definite worsening, -2 = Moderate worsening, -1 = Slight worsening, 0 = No change, 1 = Slight improvement, 2 = Moderate improvement, 3 = Definite improvement).
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
units on scale
  Baseline: OA of facial skin (n=93,97) | 5.67 (1.83) | 5.60 (1.62)
  Baseline: Fine L/W (n=93,97) | 6.51 (2.11) | 6.46 (1.89)
  Baseline: Under eye dc or bags (n=93,97) | 5.80 (2.66) | 5.82 (2.64)
  Baseline: Discoloration (n=93,97) | 5.85 (2.42) | 6.59 (2.23)
  Baseline: Complexion/Glow (n=93,97) | 5.19 (2.00) | 5.02 (1.75)
  Baseline: Smoothness (n=93,97) | 6.69 (1.92) | 6.49 (1.86)
  Improvement Week 12: OA of facial skin (n=92,96) | 0.7 (1.06) | 0.8 (0.92)
  Improvement Week 12: Fine L/W (n=92,96) | 0.4 (0.84) | 0.6 (0.89)
  Improvement Week 12: Under eye dc or bags(n=92,96) | 0.3 (0.72) | 0.3 (0.95)
  Improvement Week 12: Discoloration (n=91,95) | 0.3 (0.80) | 0.4 (1.01)
  Improvement Week 12: Complexion/Glow (n=92,96) | 0.7 (0.83) | 0.7 (0.86)
  Improvement Week 12: Smoothness (n=92,96) | 0.9 (1.01) | 1.0 (0.97)
  Improvement Week 24: OA of facial skin (n=92,96) | 0.8 (1.23) | 1.0 (1.26)
  Improvement Week 24: Fine L/W (n=92,96) | 0.6 (1.01) | 0.8 (1.18)
  Improvement Week 24: Under eye dc or bags(n=92,96) | 0.4 (0.88) | 0.5 (1.08)
  Improvement Week 24: Discoloration (n=91,93) | 0.3 (0.97) | 0.5 (1.11)
  Improvement Week 24: Complexion/Glow (n=92,96) | 0.8 (1.16) | 0.9 (1.12)
  Improvement Week 24: Smoothness (n=92,96) | 1.1 (1.22) | 1.2 (1.13)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Improvement Week 12, Overall appearance of facial skin: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.688, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.083, 95% CI 2-sided [-0.10 to 0.27]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; Improvement Week 12, Fine lines/wrinkles: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.445, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.121, 95% CI 2-sided [-0.08 to 0.33]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; Improvement Week 12, Under eye dark circles or bags: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.318, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.205, 95% CI 2-sided [0.01 to 0.40]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; Improvement Week 12, Discoloration: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.633, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.012, 95% CI 2-sided [-0.15 to 0.12]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; Improvement Week 12, Complexion/Glow: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.996, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.018, 95% CI 2-sided [-0.23 to 0.19]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; Improvement Week 12, Smoothness: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.432, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.059, 95% CI 2-sided [-0.13 to 0.25]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; Improvement Week 24, Overall appearance of facial skin: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.833, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.030, 95% CI 2-sided [-0.13 to 0.19]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; Improvement Week 24, Fine lines/wrinkles: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.171, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.226, 95% CI 2-sided [0.06 to 0.39]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; Improvement Week 24, Under eye dark circles or bags: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.796, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.020, 95% CI 2-sided [-0.16 to 0.12]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; Improvement Week 24, Discoloration: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.942, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.033, 95% CI 2-sided [-0.23 to 0.16]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; Improvement Week 24, Complexion/Glow: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.405, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.118, 95% CI 2-sided [-0.05 to 0.28]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; Improvement Week 24, Smoothness: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.687, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.061, 95% CI 2-sided [-0.14 to 0.26]

7. Secondary Outcome: Participant Improvement Assessment of Decolletage, Back of Hands and Body at Week 12 and 24
Description: Participants performed the assessment of decolletage (decolletage overall, decolletage-wrinkling/crinkling (W/C), decolletage-discoloration (DD) and back of hands (back of hands overall, back of hands (BOH) - Fine lines/wrinkles (L/W), back of hands - discoloration) and Body - Dryness (BD) Overall at baseline using a 10-point numerical scale, and at Week 12, 24 using a 7-point improvement scale. At Baseline, participants rated the Decolletage, Back of Hands and Body parameters using a 10-point scale ranging from 1 (Not noticeable) to 10 (Very noticeable). At Week 12 and 24, assessment was performed relative to Baseline using an improvement scale that ranged from -3 to 3 (where -3 = Definite worsening, -2 = Moderate worsening, -1 = Slight worsening, 0 = No change, 1 = Slight improvement, 2 = Moderate improvement, 3 = Definite improvement).
Time Frame: Baseline, Week 12, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
units on scale
  Baseline: Decolletage-Overall (n=93,97) | 5.34 (2.08) | 5.19 (1.92)
  Baseline: Decolletage-W/C (n=93,97) | 5.59 (2.35) | 5.48 (2.22)
  Baseline: Decolletage-Discoloration (n=93,97) | 5.88 (2.59) | 6.06 (2.21)
  Baseline: Back of Hands-Overall (n=93,97) | 4.89 (2.15) | 4.89 (1.98)
  Baseline: Back of Hands - Fine L/W (n=93,97) | 6.23 (2.56) | 6.53 (2.25)
  Baseline: Back of Hands - Discoloration (n=93,97) | 5.91 (2.62) | 5.83 (2.56)
  Baseline: Body - Dryness Overall (n=93,97) | 5.34 (2.23) | 5.15 (2.03)
  Improvement Week 12: Decolletage-Overall (n=92,96) | 0.3 (0.70) | 0.5 (0.75)
  Improvement Week 12: Decolletage-W/C (n=92,96) | 0.2 (0.67) | 0.4 (0.78)
  Improvement Week 12: DD (n=87,94) | 0.1 (0.57) | 0.3 (0.69)
  Improvement Week 12: BOH-Overall (n=92,96) | 0.3 (0.68) | 0.4 (0.92)
  Improvement Week 12: BOH - Fine L/W (n=92,96) | 0.2 (0.65) | 0.4 (0.90)
  Improvement Week 12: BOH - Discoloration (n=88,94) | 0.2 (0.69) | 0.3 (0.82)
  Improvement Week 12: BD Overall (n=91,96) | 0.6 (0.96) | 0.5 (1.06)
  Improvement Week 24: Decolletage-Overall (n=92,96) | 0.5 (1.00) | 0.7 (1.03)
  Improvement Week 24: Decolletage-W/C (n=92,96) | 0.5 (0.94) | 0.7 (0.98)
  Improvement Week 24: DD (n=88,91) | 0.3 (0.90) | 0.6 (1.08)
  Improvement Week 24:BOH-Overall (n=92,96) | 0.5 (0.99) | 0.7 (1.08)
  Improvement Week 24: BOH - Fine L/W (n=92,96) | 0.4 (0.93) | 0.6 (1.02)
  Improvement Week 24: BOH - Discoloration (n=91,91) | 0.3 (0.94) | 0.5 (0.97)
  Improvement Week 24: BD Overall (n=92,96) | 0.7 (1.13) | 0.7 (1.18)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Improvement Week 12, Decolletage-Overall: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.017, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.384, 95% CI 2-sided [0.23 to 0.54]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; Improvement Week 12, Decolletage-Wrinkling/crinkling: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.248, 95% CI 2-sided [0.09 to 0.40]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; Improvement Week 12, Decolletage-Discoloration: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.117, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.057, 95% CI 2-sided [-0.11 to 0.22]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; Improvement Week 12, Back of Hands-Overall: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.662, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.096, 95% CI 2-sided [-0.31 to 0.12]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; Improvement Week 12, Back of Hands - Fine lines/wrinkles: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.373, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.100, 95% CI 2-sided [-0.05 to 0.25]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; Improvement Week 12, Back of Hands - Discoloration: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.294, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.031, 95% CI 2-sided [-0.19 to 0.12]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; Improvement Week 12, Body - Dryness Overall: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.857, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.035, 95% CI 2-sided [-0.20 to 0.13]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; Improvement Week 24, Decolletage-Overall: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.088, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.206, 95% CI 2-sided [0.02 to 0.39]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; Improvement Week 24, Decolletage-Wrinkling/crinkling: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.110, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.193, 95% CI 2-sided [-0.02 to 0.41]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; Improvement Week 24, Decolletage-Discoloration: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.112, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.205, 95% CI 2-sided [0.07 to 0.34]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; Improvement Week 24, Back of Hands-Overall: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.614, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.003, 95% CI 2-sided [-0.13 to 0.13]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; Improvement Week 24, Back of Hands - Fine lines/wrinkles: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.693, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.011, 95% CI 2-sided [-0.18 to 0.16]
Statistical Analysis 13: Comparison: Placebo vs Imedeen; Improvement Week 24, Back of Hands - Discoloration: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.762, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = 0.079, 95% CI 2-sided [-0.06 to 0.22]
Statistical Analysis 14: Comparison: Placebo vs Imedeen; Improvement Week 24, Body - Dryness Overall: Analysis was performed using CMH test with modified ridit scores, controlling for Glogau Classification of Photoaging, site, and baseline; Test type: Superiority or Other; p = 0.662, Cochran-Mantel-Haenszel; Weighted Gamma Statistic = -0.013, 95% CI 2-sided [-0.16 to 0.13]

8. Secondary Outcome: Change From Baseline in Skin Hydration at Week 6, 12, 18 and 24
Description: DermaLab Combo Skin Lab with an 8-pin probe was used to measure hydration (corneometry). Hydration measurements of the left cheek, left inner arm, and left outer arm were taken (up to 3 measurement).
Time Frame: Baseline, Week 6, 12, 18, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: microsecond
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
microsecond
  Baseline: Left Cheek (n=93,97) | 231.7 (54.58) | 238.7 (69.69)
  Change at Week 6: Left Cheek (n=93,97) | -5.2 (48.13) | 1.9 (70.39)
  Change at Week 12: Left Cheek (n=87,92) | 16.7 (52.70) | 20.0 (69.01)
  Change at Week 18: Left Cheek (n=85,91) | 35.1 (47.03) | 35.5 (70.18)
  Change at Week 24: Left Cheek (n=85,91) | 33.1 (53.86) | 29.1 (71.44)
  Baseline: Left Inner Arm (n=93,97) | 150.0 (41.37) | 157.2 (52.72)
  Change at Week 6: Left Inner Arm (n=93,97) | -10.6 (48.51) | -3.7 (54.36)
  Change at Week 12: Left Inner Arm (n=87,92) | -5.2 (69.84) | 4.4 (61.24)
  Change at Week 18: Left Inner Arm (n=85,91) | 15.3 (45.69) | 15.7 (55.30)
  Change at Week 24: Left Inner Arm (n=85,91) | 15.4 (39.36) | 12.0 (53.89)
  Baseline: Left Outer Arm (n=93,97) | 120.0 (49.37) | 130.0 (61.83)
  Change at Week 6: Left Outer Arm (n=93,97) | -6.4 (42.13) | -3.5 (57.26)
  Change at Week 12: Left Outer Arm (n=87,92) | -1.5 (45.13) | 1.7 (57.49)
  Change at Week 18: Left Outer Arm (n=85,91) | 9.8 (45.27) | 14.0 (58.47)
  Change at Week 24: Left Outer Arm (n=85,91) | 9.4 (48.60) | 10.2 (50.92)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Change at Week 6, Left Cheek: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.587, ANOVA; LS Mean Difference = 3.93, 95% CI 2-sided [-10.32 to 18.18]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; Change at Week 12, Left Cheek: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.814, ANOVA; LS Mean Difference = -1.08, 95% CI 2-sided [-14.49 to 12.32]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; Change at Week 18, Left Cheek: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.453, ANOVA; LS Mean Difference = -3.57, 95% CI 2-sided [-16.14 to 8.99]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; Change at Week 24, Left Cheek: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.191, ANOVA; LS Mean Difference = -9.16, 95% CI 2-sided [-22.92 to 4.61]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; Change at Week 6, Left Inner Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.685, ANOVA; LS Mean Difference = 2.61, 95% CI 2-sided [-10.07 to 15.28]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; Change at Week 12, Left Inner Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.480, ANOVA; LS Mean Difference = 5.74, 95% CI 2-sided [-11.67 to 23.15]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; Change at Week 18, Left Inner Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.299, ANOVA; LS Mean Difference = -5.98, 95% CI 2-sided [-17.29 to 5.34]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; Change at Week 24, Left Inner Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.107, ANOVA; LS Mean Difference = -9.07, 95% CI 2-sided [-20.04 to 1.90]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; Change at Week 6, Left Outer Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.776, ANOVA; LS Mean Difference = -1.82, 95% CI 2-sided [-14.39 to 10.76]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; Change at Week 12, Left Outer Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.603, ANOVA; LS Mean Difference = -3.33, 95% CI 2-sided [-15.96 to 9.29]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; Change at Week 18, Left Outer Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.510, ANOVA; LS Mean Difference = -3.82, 95% CI 2-sided [-15.23 to 7.60]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; Change at Week 24, Left Outer Arm: Analysis was performed using ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.225, ANOVA; LS Mean Difference = -6.75, 95% CI 2-sided [-17.70 to 4.20]

9. Secondary Outcome: Change From Baseline in Trans-Epidermal Water Loss (TEWL) at Week 6, 12, 18 and 24
Description: Trans-epidermal water loss (TEWL) measurements were done using DermaLab Combo SkinLab with a cylindrical diffusion chamber (10 mm [millimeter] diameter) containing 2 combined humidity/temperature sensors to determine the amount of water vapor that moves across the stratum corneum. TEWL measurements were taken on the left cheek and the left inner and outer arm (up to 3 measurement).
Time Frame: Baseline, Week 6, 12, 18, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: gram per square meter per hour
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
gram per square meter per hour
  Baseline: Left Cheek (n=93,97) | 11.7 (5.27) | 11.0 (5.04)
  Change at Week 6: Left Cheek (n=93,97) | -0.0 (5.21) | 0.4 (4.34)
  Change at Week 12: Left Cheek (n=87,92) | 0.0 (3.72) | 0.8 (4.71)
  Change at Week 18: Left Cheek (n=85,91) | 0.2 (3.84) | 0.8 (4.35)
  Change at Week 24: Left Cheek (n=85,91) | -0.4 (4.15) | 0.4 (4.29)
  Baseline: Left Inner Arm (n=93,97) | 4.8 (2.00) | 4.4 (1.90)
  Change at Week 6: Left Inner Arm (n=93,97) | -0.3 (1.86) | -0.3 (2.46)
  Change at Week 12: Left Inner Arm (n=87,92) | -0.1 (1.79) | 0.1 (1.67)
  Change at Week 18: Left Inner Arm (n=85,91) | -0.1 (1.41) | 0.0 (1.80)
  Change at Week 24: Left Inner Arm (n=85,91) | -0.4 (1.63) | -0.2 (1.72)
  Baseline: Left Outer Arm (n=93,97) | 4.6 (1.98) | 4.1 (1.57)
  Change at Week 6: Left Outer Arm (n=93,97) | -0.2 (1.38) | -0.2 (1.81)
  Change at Week 12: Left Outer Arm (n=87,92) | -0.1 (1.53) | -0.2 (1.67)
  Change at Week 18: Left Outer Arm (n=85,91) | -0.0 (1.39) | -0.1 (1.72)
  Change at Week 24: Left Outer Arm (n=85,91) | -0.4 (1.64) | -0.4 (1.49)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.214, ANOVA; LS Mean Difference = 0.78, 95% CI 2-sided [-0.46 to 2.02]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p = 0.027, ANOVA; LS Mean Difference = 1.10, 95% CI 2-sided [0.12 to 2.09]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p = 0.049, ANOVA; LS Mean Difference = 0.99, 95% CI 2-sided [0.01 to 1.96]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p = 0.019, ANOVA; LS Mean Difference = 1.17, 95% CI 2-sided [0.20 to 2.14]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.449, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.36 to 0.80]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; p = 0.105, ANOVA; LS Mean Difference = 0.37, 95% CI 2-sided [-0.07 to 0.80]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.205, ANOVA; LS Mean Difference = 0.27, 95% CI 2-sided [-0.14 to 0.68]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; p = 0.100, ANOVA; LS Mean Difference = 0.35, 95% CI 2-sided [-0.06 to 0.77]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; p = 0.244, ANOVA; LS Mean Difference = 0.25, 95% CI 2-sided [-0.17 to 0.66]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p = 0.594, ANOVA; LS Mean Difference = 0.12, 95% CI 2-sided [-0.32 to 0.56]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; p = 0.317, ANOVA; LS Mean Difference = 0.22, 95% CI 2-sided [-0.20 to 0.63]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; [analysis description as in outcome 8, analysis 12]; Test type: Superiority or Other; p = 0.264, ANOVA; LS Mean Difference = 0.24, 95% CI 2-sided [-0.17 to 0.64]

10. Secondary Outcome: Change From Baseline in Skin Thickness at Week 6, 12,18 and 24
Description: Skin thickness was measured using the DUB Cutis (taberna pro medicum), a high frequency and high resolution diagnostic ultrasound system. Measurements were taken on the left cheek, and the left inner and outer arm (up to 3 measurement).
Time Frame: Baseline, Week 6, 12, 18, 24
Population: m-ITT population included all randomized participants who had at least 1 pre-dose and post-dose assessment value. Here "n" signifies those participants who were evaluable for this measure at specified time -points for each arm, respectively.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
micrometer
  Baseline: Left Cheek (n=93,97) | 1568.2 (234.01) | 1531.1 (243.04)
  Change at Week 6: Left Cheek (n=89,95) | 2.4 (169.50) | -33.9 (164.03)
  Change at Week 12: Left Cheek (n=87,92) | 11.3 (167.01) | -37.1 (169.86)
  Change at Week 18: Left Cheek (n=84,90) | -21.7 (173.71) | -45.8 (169.60)
  Change at Week 24: Left Cheek (n=82,90) | -55.6 (225.02) | -81.1 (230.14)
  Baseline: Left Inner Arm (n=93,96) | 1101.8 (159.25) | 1076.4 (137.32)
  Change at Week 6: Left Inner Arm (n=91,96) | 4.7 (94.41) | 3.0 (86.69)
  Change at Week 12: Left Inner Arm (n=87,91) | -11.1 (102.32) | -15.6 (92.83)
  Change at Week 18: Left Inner Arm (n=84,88) | -16.6 (117.88) | -43.2 (108.18)
  Change at Week 24: Left Inner Arm (n=82,89) | -73.2 (126.50) | -66.6 (126.87)
  Baseline: Left Outer Arm (n=93,96) | 1349.4 (191.23) | 1332.2 (169.61)
  Change at Week 6: Left Outer Arm (n=92,96) | 9.1 (106.38) | 17.0 (100.85)
  Change at Week 12: Left Outer Arm (n=87,91) | 9.5 (101.58) | 5.2 (95.81)
  Change at Week 18: Left Outer Arm (n=84,89) | -3.3 (117.71) | -23.1 (120.42)
  Change at Week 24: Left Outer Arm (n=82,89) | -55.3 (144.09) | -55.3 (135.32)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; Change at Week 6, Left Cheek: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.266, ANOVA; LS Mean Difference = -25.16, 95% CI 2-sided [-69.63 to 19.31]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; Change at Week 12, Left Cheek: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.210, ANOVA; LS Mean Difference = -28.79, 95% CI 2-sided [-73.99 to 16.41]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; Change at Week 18, Left Cheek: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.753, ANOVA; LS Mean Difference = -7.78, 95% CI 2-sided [-56.55 to 40.99]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; Change at Week 24, Left Cheek: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.632, ANOVA; LS Mean Difference = -14.90, 95% CI 2-sided [-76.32 to 46.51]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; Change at Week 6, Left Inner Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.715, ANOVA; LS Mean Difference = 4.54, 95% CI 2-sided [-19.94 to 29.01]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; Change at Week 12, Left Inner Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.648, ANOVA; LS Mean Difference = 6.35, 95% CI 2-sided [-21.04 to 33.75]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; Change at Week 18, Left Inner Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.315, ANOVA; LS Mean Difference = -16.49, 95% CI 2-sided [-48.81 to 15.83]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; Change at Week 24, Left Inner Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.402, ANOVA; LS Mean Difference = 14.42, 95% CI 2-sided [-19.50 to 48.34]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; Change at Week 6, Left Outer Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.381, ANOVA; LS Mean Difference = 12.43, 95% CI 2-sided [-15.49 to 40.35]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; Change at Week 12, Left Outer Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.916, ANOVA; LS Mean Difference = 1.49, 95% CI 2-sided [-26.44 to 29.43]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; Change at Week 18, Left Outer Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.566, ANOVA; LS Mean Difference = -9.88, 95% CI 2-sided [-43.81 to 24.05]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; Change at Week 24, Left Outer Arm: Analysis was performed using an ANOVA model with treatment, Glogau classification of photoaging, site, baseline and treatment-by-baseline interaction (if applicable) terms; Test type: Superiority or Other; p = 0.667, ANOVA; LS Mean Difference = 8.58, 95% CI 2-sided [-30.78 to 47.94]

11. Secondary Outcome: Change From Baseline in Skin Density at Week 6, 12, 18 and 24 (With 100% Calibration Mode)
Description: Skin density was measured using the DUB Cutis (taberna pro medicum), a high frequency and high resolution diagnostic ultrasound system with 100 percent (%) calibration mode. Measurements were taken on the left cheek, and the left inner and outer arm (up to 3 measurement).
Time Frame: Baseline, Week 6, 12, 18, 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Placebo | Imedeen
Number analyzed (Participants) | 93 | 97
micrometer
  Baseline: Left Cheek (n=58,59) | 10.5 (4.05) | 10.3 (3.78)
  Change at Week 6: Left Cheek (n=57,59) | -0.1 (4.43) | -0.7 (5.13)
  Change at Week 12: Left Cheek (n=54,55) | -0.1 (4.49) | -0.8 (4.34)
  Change at Week 18: Left Cheek (n=49,52) | -1.8 (5.68) | -3.3 (6.22)
  Change at Week 24: Left Cheek (n=49,53) | -2.5 (5.68) | -3.3 (5.42)
  Baseline: Left Inner Arm (n=58,58) | 28.0 (6.96) | 29.2 (8.41)
  Change at Week 6: Left Inner Arm (n=57,58) | -1.0 (10.20) | 1.2 (11.61)
  Change at Week 12: Left Inner Arm (n=54,54) | 0.3 (8.73) | -0.7 (10.05)
  Change at Week 18: Left Inner Arm (n=49,50) | -4.5 (10.73) | -4.6 (13.87)
  Change at Week 24: Left Inner Arm (n=49,52) | -6.6 (10.98) | -4.9 (11.64)
  Baseline: Left Outer Arm (n=58,58) | 19.5 (5.82) | 19.4 (6.66)
  Change at Week 6: Left Outer Arm (n=58,58) | -0.2 (7.47) | 0.0 (7.75)
  Change at Week 12: Left Outer Arm (n=54,54) | -0.5 (6.61) | -2.0 (7.93)
  Change at Week 18: Left Outer Arm (n=49,51) | -2.6 (9.01) | -3.6 (10.10)
  Change at Week 24: Left Outer Arm (n=49,52) | -4.5 (9.45) | -3.9 (9.69)
Statistical Analysis 1: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.458, ANOVA; LS Mean Difference = -0.60, 95% CI 2-sided [-2.21 to 1.00]
Statistical Analysis 2: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 2]; Test type: Superiority or Other; p = 0.497, ANOVA; LS Mean Difference = -0.53, 95% CI 2-sided [-2.07 to 1.01]
Statistical Analysis 3: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 3]; Test type: Superiority or Other; p = 0.113, ANOVA; LS Mean Difference = -1.36, 95% CI 2-sided [-3.05 to 0.33]
Statistical Analysis 4: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 4]; Test type: Superiority or Other; p = 0.708, ANOVA; LS Mean Difference = -0.34, 95% CI 2-sided [-2.11 to 1.44]
Statistical Analysis 5: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 5]; Test type: Superiority or Other; p = 0.495, ANOVA; LS Mean Difference = 1.24, 95% CI 2-sided [-2.34 to 4.82]
Statistical Analysis 6: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 6]; Test type: Superiority or Other; p = 0.243, ANOVA; LS Mean Difference = -1.85, 95% CI 2-sided [-4.96 to 1.27]
Statistical Analysis 7: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 7]; Test type: Superiority or Other; p = 0.453, ANOVA; LS Mean Difference = -1.36, 95% CI 2-sided [-4.96 to 2.23]
Statistical Analysis 8: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 8]; Test type: Superiority or Other; p = 0.745, ANOVA; LS Mean Difference = 0.55, 95% CI 2-sided [-2.79 to 3.89]
Statistical Analysis 9: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 9]; Test type: Superiority or Other; p = 0.987, ANOVA; LS Mean Difference = 0.02, 95% CI 2-sided [-2.44 to 2.48]
Statistical Analysis 10: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 10]; Test type: Superiority or Other; p = 0.218, ANOVA; LS Mean Difference = -1.42, 95% CI 2-sided [-3.69 to 0.85]
Statistical Analysis 11: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 11]; Test type: Superiority or Other; p = 0.630, ANOVA; LS Mean Difference = -0.67, 95% CI 2-sided [-3.41 to 2.08]
Statistical Analysis 12: Comparison: Placebo vs Imedeen; [analysis description as in outcome 10, analysis 12]; Test type: Superiority or Other; p = 0.576, ANOVA; LS Mean Difference = 0.81, 95% CI 2-sided [-2.06 to 3.68]

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | Imedeen
Serious Adverse Events (participants affected / at risk) | 0/95 | 2/98
Other Adverse Events (participants affected / at risk) | 24/95 | 29/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | Imedeen (N=98)
Thrombosis (Vascular disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=95) | Imedeen (N=98)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1
Gastroenteritis (Infections and infestations) | 3 | 1
Nasopharyngitis (Infections and infestations) | 3 | 8
Tooth infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 5
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.